CLINICAL TRIAL: NCT02963194
Title: Oxytocin Effects on Self and Other Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-05
Record Dates: First submitted 2016-04-15; First posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Social Behavior
Keywords: self-processing; endowment effect; neuroimage
MeSH Terms: conditions — Social Behavior | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Oxytocin (Experimental): Oxytoxin nasal spray
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Placebo nasal spray
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin
  Arms: Oxytocin
Drug: Placebo
  Arms: Placebo

SUMMARY:
To determine whether the neuropeptide oxytocin (OXT) influences self-processing by investigating whether it increases the endowment effect in relation to both self and others.

DETAILED DESCRIPTION:
In a double-blind, between- subject placebo (PLC) controlled design, investigator aimed to measure the effect of intranasal OXT on the endowment effect. All subjects completed a range of questionnaires measuring personality and affective traits and levels of anxiety before self-administration: Positive and Negative Affect Schedule (PANAS) , State-Trait Anxiety Inventory (STAI) , Beck Depression Inventory (BDI), self-esteem scale (SES). Subjects were asked to decide whether to buy or sell their own or others' (their mothers'/ fathers'/ classmate'/ strangers') possessions at various prices. Indifference point and brain activation were inluded into analysis as dependent variables.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* history of head injury;
* claustrophobia;
* medical or psychiatric illness.

Ages: 18 Years to 27 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Compared the indifference point between buy and sell conditions during the price phase and the specific brain region activation between oxytocin and placebo groups | 1 hour
  Indifference point is the gap between willingness to accept and willingness to pay ;focus on the specfic brain region relasted to self-processing, such as medial prefrontal cortex, precuneus, posterior cingulate cortex, ventral striatum.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, Dr., Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- School of Life Science and Technology, University of Electronic Science and Technology, Chengdu, Sichuan, China